CLINICAL TRIAL: NCT06438666
Title: A Quasi Experimental Study About the Effects Obtained at Manual Function After Applying Anodic Transcranial Direct Current Stimulation in Children With Spastic Hemiparetic Cerebral Palsy
Brief Title: Effects Obtained at Manual Function After Applying Anodic Transcranial Direct Current Stimulation (tCDS) in Children With Spastic Hemiparetic Cerebral Palsy
Acronym: PeditCDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Jorge Manuel Góngora Rodríguez (Unknown)
Responsible Party: Principal Investigator, Rocío Martín Valero, Director, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tDCS_2024UMA
Record Dates: First submitted 2024-05-23; First posted 2024-06-03 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hemiparetic Cerebral Palsy
Keywords: Cerebral Palsy; Transcranial Direct Current Stimulation; Upper Limb
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: 20 participants between 14-18 years old will receive 4 sessions of anodic transcranial direct current stimulation. The results will be measured before and after the 4 sessions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with spactic hemiparetic cerebral palsy (Experimental): A group of children with spastic hemiparetic cerebral palsy will be treated with anodic transcranial direct currents.
  Interventions: Device: Anodic Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Anodic Transcranial Direct Current Stimulation — This study will apply the anodic transcranial direct current stimulation over 20 children between 14-18 years old. The protocol that it will follow is the next one: 3 days to value the outcome measures, 4 days (1 sessions per day of 17 minutes and 30 seconds) to apply the protocol of anodic transcranial direct current stimulation (0,6 mA of intensity). It will use the EPTE V07 Bipolar System by IONCLINICS ®; 3 days to value the outcome measures studying the effects produced at the affected upper limb. Another evaluation will be realized 3 weeks after the last sessions of anodic transcranial direct current stimulation to know if the effects obtained last at medium-long term.

SUMMARY:
Spastic Hemiparetic Cerebral Palsy (SHCP) uses to limit the manual function. Using anodic transcranial direct current stimulation, it is possible to activate certain cerebral areas depending on where the electrodes are. This study will use this kind of stimulation on the contralateral primary motor cortex of the affected upper limb and analyze the effects.

DETAILED DESCRIPTION:
It has been designed a single-arm prospective longitudinal quasi-experimental pilot clinical study following the SPIRIT 2013 statement. It will value the time that the children spend doing the bimanual activities described by the Children's Hand-Use Experience Questionnaire (CHEQ), it will also value the subjective experience doing those activities; it will analyze the active movement (Fugl-Meyer for upper limb), spasticity (modified Ashworth), manual strength (dynamometry) and the recruitment improvement (surface electromyography) too.

This study will apply the anodic transcranial direct current stimulation over 20 children between 14-18 years old. The protocol that it will follow is the next one: 3 days to value the outcome measures, 4 days (1 session per day of 17 minutes and 30 seconds) to apply the protocol of anodic transcranial direct current stimulation (0,6 mA of intensity). It will use the EPTE V07 Bipolar System by IONCLINICS ®; 3 days to value the outcome measures studying the effects produced at the affected upper limb. Another evaluation will be realized 3 weeks after the last session of anodic transcranial direct current stimulation to know if the effects obtained last at medium-long term.

ELIGIBILITY:
Inclusion Criteria:

* Children between 14-18 years old.
* Children with spastic hemiparetic cerebral palsy diagnosis.
* Children with a cognitive level high enough to understand and to do the activities to value them.
* Children hemodynamically stable.
* Children forming part of levels II-IV of the Manual Ability Classification System (MACS).

Exclusion Criteria:

* Children with defibrillator.
* Children with pacemaker.
* Children with cerebral stimulator.
* Children with intracranial metallic implants.
* Children with opened cranial after clambering.
* Children that receive another treatment (pharmacological or physiotherapical) that could interfere or disrupt the results.
* Another circumstance where the electrotherapy treatment is contraindicated.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-12-23 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Changes in the timing that children use to complete the 29 items of the Children's Hand-Use Experience Questionnaire (CHEQ). | Baseline, after 4 days (after de foruth sessions planned) and 3 weeks later
  CHEQ is a questionnaire analyze the time it takes the children (between 6-18 years old) to do 29 functional activities; it also values the subjective experience of the children doing theses activities. It has a punctuation that goes from 1 to 4 (the maximum score is 348). If the score is higher, it means that the children's status is better.

SECONDARY OUTCOMES:
Changes at the spasticity | Baseline, after 4 days (after the fourth sessions planned) and 3 weeks later
  Ashworth modified scale is a scale that values the spasticity. It has a punctuation that goes from 0 to 4. If the score is higher, it means that the spasticity is worse.
Changes at the active movement | Baseline, after 4 days (after the fourth sessions planned) and 3 weeks later
  Fugl-Meyer scale for upper limb Is a scale that values the active movement, the sensibility, joints pain and passive movement of the upper limb. It has a punctuation that goes from 0 to 2 (the maximun score is 126). If the score is higher, it means that all it values are fine.
Changes at the manual strength | Baseline, after 4 days (after the fourth sessions planned) and 3 weeks later
  Dynamometry is a test that values the hand strength.
Changes at the recruitment of the motor units. | Baseline, after 4 days (after the fourth sessions planned) and 3 weeks later
  Surface electromyography is a test that values the improvement in the recruitment of the motor units.

CONTACTS AND LOCATIONS:
Locations (1):
- Rocío Martín Valero, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mediline Plus — https://medlineplus.gov/spanish/
- See also: Brain Stimulation Therapies — https://www.nimh.nih.gov/health/topics/brain-stimulation-therapies/brain-stimulation-therapies